CLINICAL TRIAL: NCT03967444
Title: Post Marketing Study to Evaluate Lip Augmentation & Satisfaction With Restylane Kysse
Brief Title: Study to Evaluate Satisfaction After Treatment With Kysse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05DF1807
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Results first posted 2021-03-01 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2021-02

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restylane Kysse (Other): Hyaluronic acid
  Interventions: Device: Hyaluronic acid
- Restylane Kysse with other HA (Other): Hyaluronic acid
  Interventions: Device: Hyaluronic acid

INTERVENTIONS:
Device: Hyaluronic acid — Injectable gel for lip augmentation
  Other Names: Restylane Kysse
  Arms: Restylane Kysse
Device: Hyaluronic acid — Injectable gel. Lip Augmentation and other wrinkles/folds
  Other Names: Restylane Kysse with other Restylane products
  Arms: Restylane Kysse with other HA

SUMMARY:
Open-label, phase IV, post-marketing study to evaluate aesthetic improvement and satisfaction after treatment with Kysse.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent to participate in the study
* Adult women and men who intend to undergo lip augmentation

Exclusion Criteria:

* Subjects presenting with known allergy to HA (hyaluronic acid) filler or amide local anesthetics
* Subjects with a previous implant other than HA in or near the intended treatment site
* Participation in any other clinical study within three (3) months before treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Galderma R&D
Locations (2):
- Canada (2):
  - Galderma Study Site, Montreal
  - Galderma Study Site, Toronto

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restylane Kysse | Restylane Kysse With Other HA
Started | 19 | 40
Completed | 18 | 38
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restylane Kysse | Restylane Kysse With Other HA | Total
Number analyzed (Participants) | 19 | 40 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 38 | 56
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (13.26) | 50.9 (10.53) | 46.2 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 38 | 56
  Male | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 1 | 2
  Race: White | 17 | 36 | 53
  Race: Other | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 19 | 40 | 59

OUTCOME MEASURES:

1. Primary Outcome: Assess Treatment With Restylane Kysse Using GAIS
Description: The 5-grade Global Aesthetic Improvement Scale (GAIS) assess the appearance of the lips compared to pre-treatment. The rating is very much improved, much improved, improved, no change, or worse. Responders are those with a rating of at least improved.
Time Frame: 8 weeks after last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Kysse | Restylane Kysse With Other HA
Number analyzed (Participants) | 18 | 38
Participants | 18 | 38

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Restylane Kysse | Restylane Kysse With Other HA
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/40
Other Adverse Events (participants affected / at risk) | 10/19 | 25/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Kysse (N=19) | Restylane Kysse With Other HA (N=40)
Implant Site Bruising (General disorders) | 6 (8) | 17 (31)
Implant Site Pain (General disorders) | 6 (12) | 14 (41)
Implant Site Oedema (General disorders) | 7 (15) | 9 (23)
Impalnt site erythema (General disorders) | 3 (5) | 10 (21)
Implant Site Swelling (General disorders) | 1 (1) | 3 (3)
Implant Site Reaction (General disorders) | 0 (0) | 1 (1)
Implant Site Dysaesthesia (General disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Animal Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT03967444/Prot_001.pdf
  • Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT03967444/SAP_000.pdf